CLINICAL TRIAL: NCT05155397
Title: The Dortmund Vital Study: Impact of Biological and Lifestyle Factors on Cognitive Performace and Work Ability Across the Lifespan. An Interdisciplinary, Cross-sectional and Longitudinal Study
Brief Title: The Dortmund Vital Study: Impact of Biological and Lifestyle Factors on Cognitive Performace and Work Ability
Acronym: DVS
Status: Active, not recruiting | Type: Observational
Sponsor: Technical University of Dortmund (Other)
Responsible Party: Sponsor
Other Study IDs: A93-3
Record Dates: First submitted 2021-11-16; First posted 2021-12-13 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Age-related Cognitive Decline
Keywords: Cognitive Ageing; Occupational Health; Neuropsychology; Metabolism; Cardiovascular System; Behavioral Genetics; Immunology; EEG; MRI; psychoneuroendocrinology; Infectious diseases; Cognitive Neuroscience
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral venous blood, serum, urine, hair samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of the Dortmund Vital Study is to validate previous hypotheses and to generate and validate new hypotheses about the relationship of ageing, working conditions, genetic makeup, stress, metabolic functions, cardiovascular system, immune system, and mental performance over the lifespan with a focus on healthy working adults. The Dortmund Vital Study is a multidisciplinary longitudinal study involving the Departments of Ergonomics, Immunology, Psychology and Neurosciences, and Toxicology of the Leibniz Research Centre for Working Environment and Human Factors at the TU Dortmund (IfADo) in Dortmund, Germany, as well as several national and international cooperation partners.

DETAILED DESCRIPTION:
The Dortmund Vital Study is designed as a combined cross-sectional and longitudinal study. About 600 subjects aged between 20 and 70 years will participate. A wide range of demographic, psychological, behavioral, sensory, cardiovascular, biochemical, immunological and biochemical data, a comprehensive EEG-based cognitive test battery as well as structural and functional magnetic resonance imaging (MRI) have been included in the study. Specifically, parameters obtained by MRI and EEG-related measures can be evaluated as a function of polygenic scores, metabolic products, concentration of immune cells, immune age and infections, such as Toxoplasmosis or COVID-19 that are largely unexplored. The same is true for environmental and lifestyle factors that impact on brain activity and behavior.

The initial testing has been conducted between 2016 and 2021 and will be repeated every five years (three follow-up measures until 2035).

The study will shed light on sources of large inter-individual differences in cognitive functioning with increasing age and reveal biological and lifestyle markers contributing to work ability, longevity and healthy aging on the one hand, and on risk factors for cognitive decline, mild cognitive impairment or even dementia on the other.

ELIGIBILITY:
Inclusion Criteria:

* Blood thinners
* Hormones
* Antihypertensives
* Cholesterol reducers
* Normal or corrected-to-normal vision and hearing
* Fulfill standard inclusion criteria for MRI measurements
* Sufficient language skills

Exclusion Criteria:

* Dementia
* Parkinsonism
* Stroke
* Cardiovascular diseases
* Bleeding tendency
* Oncological diseases
* Schizophrenia
* Obsessive-compulsive disorder
* Anxiety disorders
* Severe depression
* Head injuries
* Head surgery
* Head implants
* Eye diseases (cataract, glaucoma, blindness)
* Accidents that limit physical fitness and mobility
* Psychotropic drugs
* Neuroleptics

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy individuals from the general population.
Sampling Method: Non-Probability Sample
Enrollment: 627 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2035-12 (Estimated); Study Completion 2037-12 (Estimated)

PRIMARY OUTCOMES:
Change in performance on global cognitive composite score assessed by neuropsychological tests | Baseline and 5, 10, 15 years
  Change in performance on global cognitive composite score based on measures from neuropsychological tests: Digit-Span forward and backward, semantic memory in written and spoken versions (Word-Fluency), selective attention and attentional endurance (D2-R), crystallized intelligence (Multiple Choice Vocabulary Test), general cognitive status (Mini-Mental-State-Examination; MMSE), different aspects of verbal memory like learning performance and retrieval (Verbal Learning and Memory Tests; VLMT), psychomotor performance and speed of processing (Digit-Symbol-Test), interference control and inhibition (Stroop Test), task switching (Trail-Making-Test; TMT-A and TMT-B), two subtests from the performance testing system measuring logical reasoning and spatial rotation, and fluid intelligence assessed by Raven's Progressive Matrices.
Change in attentional performance and perceptual control as assessed by a computerized Bar Task | Baseline and 5, 10, 15 years
  Changes in behavioral (speed and accuracy) and electroencephalogram (EEG) data in attentional performance and perceptual control assessed by the Bar Task.
Change in vigilance control as assessed by a computerized Psychomotor Vigilance Test | Baseline and 5, 10, 15 years
  Changes in behavioral (speed and accuracy) and electroencephalogram (EEG) data in a Psychomotor Vigilance Test.
Change in stimulus-response compatibility and conflict processing assessed by the computerized Simon Task | Baseline and 5, 10, 15 years
  Changes in behavioral (speed and accuracy) and electroencephalogram (EEG) data in the Simon task.
Change in updating and strategy learning assessed by the computerized AX-CPT Task | Baseline and 5, 10, 15 years
  Changes in behavioral (speed and accuracy) and electroencephalogram (EEG) data in the AX-CPT task.
Change in speech understanding and auditory distractibility assessed by computerized Speech-In-Noise perception task | Baseline and 5, 10, 15 years
  Changes in behavioral (speed and accuracy) and electroencephalogram (EEG) data in the Speech-in-noise perception task.
Change in working memory assessed by the computerized N-back Task | Baseline and 5, 10, 15 years
  Changes in behavioral (speed and accuracy) and electroencephalogram (EEG) data in the N-back task.
Change in cue and memory-based task switching assessed by the computerized Task Switching Paradigm | Baseline and 5, 10, 15 years
  Changes in behavioral (speed and accuracy) and electroencephalogram (EEG) data in the cue- and memory based task switching.
Change in auditive attention and distractibility assessed by the computerized Auditory Distraction Task | Baseline and 5, 10, 15 years
  Changes in behavioral (speed and accuracy) and electroencephalogram (EEG) data in the Auditory Distraction Task.
Change in susceptibility to interference and the capacity to inhibit irrelevant stimuli assessed by the computerized Stroop Task | Baseline and 5, 10, 15 years
  Changes in behavioral (speed and accuracy) and electroencephalogram (EEG) data in the Stroop Task.
Change in inhibitory control of prepotent responses assessed by the computerized Go/NoGo Task | Baseline and 5, 10, 15 years
  Changes in behavioral (speed and accuracy) and electroencephalogram (EEG) data in the Go/NoGo Task.
Change in spatial selective attention assessed by the computerized Visual Search Task | Baseline and 5, 10, 15 years
  Changes in behavioral (speed and accuracy) and electroencephalogram (EEG) data in the Visual Search Task.
Change in Work Ability Index | Baseline and 5, 10, 15 years
  Change in work ability assessed by Work Ability Index (WAI). WAI assess physical and psychological risks to avoid work-related disabilities and early retirement. The index is determined by the employees' answers related to work demands, individual health status and physical and psychological capacities. The total score of WAI is calculated by summing up scores of seven dimensions. The work ability ranged between 7 (insufficient) and 49 points (best work ability).

SECONDARY OUTCOMES:
Change in resting state EEG activity | baseline and 5, 10, 15 years
  Change in resting state EEG activity measured for 2 minutes with eyes open, and 2 minutes with eyes closed.
Change in brain function MRI | 5, 10, 15 years
  Changes in functional magnetic resonance imaging assessed by resting state MRI.
Change in brain structure MRI | 5, 10, 15 years
  Changes in structural resonance imaging assessed by multi-shell diffusion-weighted imaging (DWI).
Change in Depressive Symptoms | Baseline and 5, 10, 15 years
  Change in total score using the Becks Depression Inventory (BDI).
Change in Burnout Symptoms | Baseline and 5, 10, 15 years
  Change in total score using the Maslach Burnout Inventory (MBI-D) with 6-point Likert-type scale ranging from 1 (never) to 6 (always), total scores: 14 - 84. Higher scores indicate more severe symptoms.
Change in Burnout Symptoms | Baseline and 5, 10, 15 years
  Change in total score using the Oldenburg Burnout Inventory (OLBI). 4-point Likert-type scale ranging from 1 (strongly agree) to 4 (strongly disagree), total scores: 8 - 32. Higher scores indicate more severe symptoms.
Change in Psychosocial Stress Symptoms | Baseline and 5, 10, 15 years
  Change in total score using the Psychosocial Stress Questionnaire (PSQ-20).
Change in Chronic Stress Symptoms | Baseline and 5, 10, 15 years
  Change in chronic stress symptoms assessed by the Trier Inventory of Chronic Stress (TICS), consisting of several dimensions: Work Overload, Social Overload, Pressure to Perform, Work Discontent, Demands from work, Lack of Social Recognition, Social Tensions, Social Isolation, Chronic Worrying, and a 12 Item Screening-Scale (SSCS) that provides a score for general stress.
Change in Psychosocial Work Demands | 5, 10, 15 years
  Change in total score in the Copenhagen Psychosocial Questionnaire (COPSOQ III) that consists of several dimensions: cognitive and physical demands at work, job control, influence at work, developmental possibilities, interpersonal relations, leadership, and strain.
Change in Self-Control at work | Baseline and 5, 10, 15 years
  Change of the psychosocial demands at work assessed by the scale Self-Control at Work.
Change in Cognitive Failures in the Daily Life | Baseline and 5, 10, 15 years
  Change in cognitive failures in daily life assessed by the Cognitive Failure Questionnaire (CFQ).
Change in Positive and Negative Affect | Baseline and 5, 10, 15 years
  Change in scores of positive and negative affect. The Positive and Negative Affect Schedule (PANAS) is a self-report questionnaire that consists of two 10-item scales to measure both positive and negative affect.
Change in Quality of Life | Baseline and 5, 10, 15 years
  Change in total score of the quality of life questionnaire (WHOQoL-BREF), consisting of dimensions: physical, psychological, social, environmental, and global quality of life.
Change in sociodemographic parameters | Baseline and 5, 10, 15 years
  Change in different sociodemographic aspects like marital status, occupational status, nutrition, leisure activities, alcohol drinking, frequency of social contacts, using of electronic media etc. Qualitative data will be categorized.
Change in self-reported physical activity | Baseline and 5, 10, 15 years
  Change of the self-reported physical activity (Lüdenscheid Physical Activity Questionnaire) in minutes per week.
Change in lateralization and motor functions | Baseline and 5, 10, 15 years
  Change in total score of the Perdue Pegboard Test, assessing lateralization and motor functions.
Change of cytokines concentration in serum | Baseline and 5, 10, 15 years
  Change of concentration of cytokines in serum (pg/ml): (IL-1b, IFN-alpha, IFN-gamma, TNF-alpha, MCP-1, IL-6, IL-8, IL-10, IL-12p70, IL-17A, IL-18, IL-23, IL-33).
Change of functional activiy of T cells and Natural Killer cells | Baseline and 5, 10, 15 years
  Change of functional activities of T cells and natural killer cells in %.
Change of peripheral blood mononuclear cells concentration | Baseline and 5, 10, 15 years
  Change of peripheral blood mononuclear cells concentration (pg/ml): (PBMC; CD14 positive monocytes).
Change in physical performance | Baseline and 5, 10, 15 years
  Change of physical fitness assessed by bicycle ergometer and a physical work capacity cycle test (PWC-130) to predict the absolute power output (in Watt) at a projected heart rate of 130 beats per minute. A relative power output is calculated by the power-to-weight ratio (Watt/kg).
Change in cardiovascular parameters | Baseline and 5, 10, 15 years
  Diastolic and systolic blood pressure (mm/Hg) and pulse (bpm) measured during rest and during cycle ergometry.
Change in electrocardiography | Baseline and 5, 10, 15 years
  Change in electrocardiogram (ECG) measured during rest and during cycle ergometry.
Change in antibody concentrations of Toxoplasma gondii in serum | Baseline and 5, 10, 15 years
  Change of concentration of Toxoplasma gondii IgG antibodies (pg/ml) in serum to assess the severity of latent toxoplasmosis infection.
Change in antibody concentrations of COVID-19 in serum | 5, 10, 15 years
  Concentration of COVID-19 antibodies (pg/ml) in serum to assess the intensity of immunological response to potential SARC-CoV-2 infection or response to vaccination.
Change in metabolic parameters in blood | Baseline and 5, 10, 15 years
  Change in metabolic parameters in serum (pg/ml): concentration of ammonia, leucocytes, erythrocytes, hematocrit, monocytes, creatinine, lymphocytes, cell volume, thrombocytes, triglycerides, cholesterol, high- and low-density lipoprotein cholesterol, glycosylated hemoglobin, glucose, C-reactive protein and creatinine are measured in venous blood.
Change of metabolic parameters in urine | Baseline and 5, 10, 15 years
  Change in metabolic parameters in urine (pg/ml): concentartion of creatinine and calcium oxalate.
Change of endocrine parameter | Baseline and 5, 10, 15 years
  Change of hair cortisol concentration (pg/mg) as an index of long-term stress.

OTHER OUTCOMES:
Genetic parameters (Single Nucleotide Polymorphisms; SNP) | Baseline
  A number of genetic polymorphisms coding common homozygotes, heterozygotes and rare homozygotes variants were selected which are potentially related to structure and function of the central nervous system. Blood samples were used for the DNA-genotyping of: Apo-E2, E3, E4 (rs7412, rs429358), BDNF Val66Met (rs6265), COMT-1 (rs4633), COMT-2 Val158Met (rs4680), DRD2 (rs6277, DRD1-48A/G (rs4532), CHRNA6-1 (rs1072003), CHRNA6-3 (rs2304297), CHRNB3-1 (rs13280604), CHRNB3-2 (rs4950), GPCPD1 (EDI3) (rs)6116869), GRIN2A (rs1969060), GRIN2A (rs8057394), GRIN2B (rs890), IL-1beta (rs16944), IL-6 (rs1800795), IL-12A (rs568408), TNF-alpha (rs1800629).
Change in visual acuity | Baseline and 5, 10, 15 years
  Change in visual acuity assessed by Vistec's Optovist according to DIN 58220-3 "Visual acuity testing - Part 3: Test for use in expertise" for far vision with the right and left eye separately (monocular) and with both eyes together (binocular), and if available with correction for distance (glasses for far vision). The "inclined optometer" is used to determine the zones of sufficient vision binocular at horizontal gaze inclination. For this, the near and far points are obtained, if available with distance correction (glasses for far vision).
Change in auditory acuity | Baseline and 5, 10, 15 years
  Change in auditory acuity evaluated by audiometry. Audiometric thresholds are tested for ten pure-tone frequencies (125, 250, 500, 750, 1000, 2000, 3000, 4000, 6000, 8000 Hz) for the left and right ears separately.
Change in Body Mass Index | Baseline and 5, 10, 15 years
  Height (m) and weight (kg) are measured to compute the Body Mass Index (BMI in kg/m^2).
Change in Waist-To-Hip ratio | Baseline and 5, 10, 15 years
  Waist- and hip measurements (cm) are measured to compute the waist-to-hip ratio.
Personality traits | Baseline
  Personality traits are evaluated by the Big-Five-Factor inventory (NEO-FFI), assessing the personality dimensions: neuroticism, extraversion, openness, agreeableness, and conscientiousness. Grit personality trait are assessed by the GRID scale and the self-control by the general self-control scale.
Stress reactivity | Baseline
  Subjective stress reactivity are assessed by the Perceived Stress Reactivity Scale (PSRS).
Chronotype | Baseline
  The chronotype assessing the morning or evening type is evaluated by (D-MEQ).
Handedness | Baseline
  Handedness is evaluated by Handedness Edinburgh Inventory.
Traumatic Experiences During Childhood | Baseline
  Traumatic experiences during childhood are assessed to evaluate stress reactivity in the adult life.
Sociodemographic characteristics | Baseline
  Sociodemographic characteristics like education, history of physical activity, marital status, children etc. were obtained. Qualitative data are categorized.
Experiences with COVID-19 pandemic | 5, 10, 15 years
  Questionnaire addressing COVID-19-specific experience with the pandemic and the consequences of a COVID-19 infection (if applicable).

CONTACTS AND LOCATIONS:
Overall Officials: Edmund Wascher, PhD, Study Director — Leibniz Research Centre for Working Environment and Human Factors at the TU Dortmund (IfADo)
Locations (1):
- Technical University of Dortmund, Leibniz Research Centre for Working Environment and Human Factors, Dortmund, Germany

IPD SHARING:
Plan to Share IPD: Yes
After primary analyses and publication of the main results the data and the scripts used for data analyses will be made available in repositories for secondary analyses. The transfer agreement will be prepared by the coordinators of the Dortmund Vital Study in consultation with the IfADo Research Data Management Unit.
Supporting Information: Study Protocol, Analytic Code
Time Frame: After primary analyses and publication of the main results.
Access Criteria: In order to access the data, scientists from IfADo, as well as external cooperation partners who plan to analyze data from the Dortmund Vital Study fill in a proposal form that includes a short description of the project and the respective hypotheses, the responsible persons, cooperation partners, data usage and analysis strategy. The requested research data will be made available in an anonymized form after consultation with the scientists responsible for the data. Responsible persons include project managers and coordinators of the Dortmund Vital Study in consultation with the IfADo Research Data Management Unit.

REFERENCES:
- [Background] Gajewski PD, Getzmann S, Brode P, Burke M, Cadenas C, Capellino S, Claus M, Genc E, Golka K, Hengstler JG, Kleinsorge T, Marchan R, Nitsche MA, Reinders J, van Thriel C, Watzl C, Wascher E. Impact of Biological and Lifestyle Factors on Cognitive Aging and Work Ability in the Dortmund Vital Study: Protocol of an Interdisciplinary, Cross-sectional, and Longitudinal Study. JMIR Res Protoc. 2022 Mar 14;11(3):e32352. doi: 10.2196/32352. PMID 35285810
- [Result] Kleinert T, Nash K, Koenig T, Wascher E. Correction: Normative Intercorrelations between EEG Microstate Characteristics. Brain Topogr. 2024 Mar;37(2):270. doi: 10.1007/s10548-023-01012-4. No abstract available. PMID 37861818
- [Result] Kleinert T, Nash K, Koenig T, Wascher E. Normative Intercorrelations Between EEG Microstate Characteristics. Brain Topogr. 2024 Mar;37(2):265-269. doi: 10.1007/s10548-023-00988-3. Epub 2023 Jul 14. PMID 37450085
- [Result] Kleinert T, Koenig T, Nash K, Wascher E. On the Reliability of the EEG Microstate Approach. Brain Topogr. 2024 Mar;37(2):271-286. doi: 10.1007/s10548-023-00982-9. Epub 2023 Jul 6. PMID 37410275
- [Result] Getzmann S, Arnau S, Gajewski PD, Wascher E. Auditory distraction, time perception, and the role of age: ERP evidence from a large cohort study. Neurobiol Aging. 2024 Dec;144:114-126. doi: 10.1016/j.neurobiolaging.2024.09.012. Epub 2024 Sep 20. PMID 39316947
- [Result] Getzmann S, Gajewski PD, Schneider D, Wascher E. Resting-state EEG data before and after cognitive activity across the adult lifespan and a 5-year follow-up. Sci Data. 2024 Sep 10;11(1):988. doi: 10.1038/s41597-024-03797-w. PMID 39256413
- [Result] Mundorf A, Getzmann S, Gajewski PD, Larra MF, Wascher E, Genc E, Ocklenburg S. Phenotyping in clinical laterality research: a comparison of commonly used methods to determine mixed-handedness and ambidexterity. Laterality. 2024 May;29(3):331-349. doi: 10.1080/1357650X.2024.2370871. Epub 2024 Jul 5. PMID 38968414
- [Result] Larra MF, Gajewski PD, Getzmann S, Wascher E, Metzler Y. Stress from early life to adulthood: Is there a protective role of cognitive control? Brain Cogn. 2024 Aug;178:106165. doi: 10.1016/j.bandc.2024.106165. Epub 2024 May 16. PMID 38759431
- [Result] Getzmann S, Golka K, Brode P, Reinders J, Kadhum T, Hengstler JG, Wascher E, Gajewski PD. Chronic Toxoplasma gondii Infection Modulates Hearing Ability across the Adult Life Span. Life (Basel). 2024 Jan 29;14(2):194. doi: 10.3390/life14020194. PMID 38398703
- [Result] Brode P, Claus M, Gajewski PD, Getzmann S, Wascher E, Watzl C. From Immunosenescence to Aging Types-Establishing Reference Intervals for Immune Age Biomarkers by Centile Estimation. Int J Mol Sci. 2023 Aug 24;24(17):13186. doi: 10.3390/ijms241713186. PMID 37685992
- [Result] Gajewski PD, Golka K, Hengstler JG, Kadhum T, Digutsch J, Genc E, Wascher E, Getzmann S. Does physical fitness affect cognitive functions differently across adulthood? An advantage of being older. Front Psychol. 2023 Jun 16;14:1134770. doi: 10.3389/fpsyg.2023.1134770. eCollection 2023. PMID 37397318
- [Result] Rieker JA, Gajewski PD, Reales JM, Ballesteros S, Golka K, Hengstler JG, Wascher E, Getzmann S. The impact of physical fitness, social life, and cognitive functions on work ability in middle-aged and older adults. Int Arch Occup Environ Health. 2023 May;96(4):507-520. doi: 10.1007/s00420-022-01943-8. Epub 2022 Dec 16. PMID 36525080
- [Result] Akan O, Bierbrauer A, Kunz L, Gajewski PD, Getzmann S, Hengstler JG, Wascher E, Axmacher N, Wolf OT. Chronic stress is associated with specific path integration deficits. Behav Brain Res. 2023 Mar 28;442:114305. doi: 10.1016/j.bbr.2023.114305. Epub 2023 Jan 20. PMID 36682499
- [Result] Getzmann S, Arnau S, Gajewski PD, Wascher E. When long appears short: Effects of auditory distraction on event-related potential correlates of time perception. Eur J Neurosci. 2022 Jan;55(1):121-137. doi: 10.1111/ejn.15553. Epub 2021 Dec 14. PMID 34859527
- [Result] Getzmann S, Schneider D, Wascher E. Selective spatial attention in lateralized multi-talker speech perception: EEG correlates and the role of age. Neurobiol Aging. 2023 Jun;126:1-13. doi: 10.1016/j.neurobiolaging.2023.02.003. Epub 2023 Feb 14. PMID 36881943
- [Result] Wascher E, Sharifian F, Gutberlet M, Schneider D, Getzmann S, Arnau S. Mental chronometry in big noisy data. PLoS One. 2022 Jun 8;17(6):e0268916. doi: 10.1371/journal.pone.0268916. eCollection 2022. PMID 35675345
- [Result] Sharifian F, Schneider D, Arnau S, Wascher E. Decoding of cognitive processes involved in the continuous performance task. Int J Psychophysiol. 2021 Sep;167:57-68. doi: 10.1016/j.ijpsycho.2021.06.012. Epub 2021 Jul 1. PMID 34216693
- [Result] Getzmann S, Digutsch J, Kleinsorge T. COVID-19 Pandemic and Personality: Agreeable People Are More Stressed by the Feeling of Missing. Int J Environ Res Public Health. 2021 Oct 13;18(20):10759. doi: 10.3390/ijerph182010759. PMID 34682500
- [Result] Metzen D, Genc E, Getzmann S, Larra MF, Wascher E, Ocklenburg S. Frontal and parietal EEG alpha asymmetry: a large-scale investigation of short-term reliability on distinct EEG systems. Brain Struct Funct. 2022 Mar;227(2):725-740. doi: 10.1007/s00429-021-02399-1. Epub 2021 Oct 21. PMID 34676455
- [Result] Bierbrauer A, Kunz L, Gomes CA, Luhmann M, Deuker L, Getzmann S, Wascher E, Gajewski PD, Hengstler JG, Fernandez-Alvarez M, Atienza M, Cammisuli DM, Bonatti F, Pruneti C, Percesepe A, Bellaali Y, Hanseeuw B, Strange BA, Cantero JL, Axmacher N. Unmasking selective path integration deficits in Alzheimer's disease risk carriers. Sci Adv. 2020 Aug 28;6(35):eaba1394. doi: 10.1126/sciadv.aba1394. eCollection 2020 Aug. PMID 32923622
- [Result] Gajewski PD, Hanisch E, Falkenstein M, Thones S, Wascher E. What Does the n-Back Task Measure as We Get Older? Relations Between Working-Memory Measures and Other Cognitive Functions Across the Lifespan. Front Psychol. 2018 Nov 26;9:2208. doi: 10.3389/fpsyg.2018.02208. eCollection 2018. PMID 30534095
- [Result] Brode P, Claus M, Gajewski PD, Getzmann S, Golka K, Hengstler JG, Wascher E, Watzl C. Calibrating a Comprehensive Immune Age Metric to Analyze the Cross Sectional Age-Related Decline in Cardiorespiratory Fitness. Biology (Basel). 2022 Oct 27;11(11):1576. doi: 10.3390/biology11111576. PMID 36358277
- [Result] Mundorf A, Getzmann S, Gajewski PD, Larra MF, Wascher E, Ocklenburg S. Stress exposure, hand preference, and hand skill: A deep phenotyping approach. Laterality. 2023 Mar-May;28(2-3):209-237. doi: 10.1080/1357650X.2023.2204551. Epub 2023 Apr 26. PMID 37099727
- [Result] Gajewski PD, Rieker JA, Athanassiou G, Brode P, Claus M, Golka K, Hengstler JG, Kleinsorge T, Nitsche MA, Reinders J, Tisch A, Watzl C, Wascher E, Getzmann S. A Systematic Analysis of Biological, Sociodemographic, Psychosocial, and Lifestyle Factors Contributing to Work Ability Across the Working Life Span: Cross-sectional Study. JMIR Form Res. 2023 May 19;7:e40818. doi: 10.2196/40818. PMID 37204831
- [Derived] Brode P, Claus M, Getzmann S, Golka K, Hengstler JG, Reinders J, Wascher E, Watzl C, Gajewski PD. Latent Toxoplasma gondii Infection Does Not Modulate Immune Aging in a Cross-Sectional Working-Age Population Study. Biomolecules. 2025 Dec 30;16(1):55. doi: 10.3390/biom16010055. PMID 41594595
- [Derived] Engler R, Stammen C, Arnau S, Schneider Penate J, Metzen D, Digutsch J, Gajewski PD, Getzmann S, Fraenz C, Reinders J, Voelkle MC, Streit F, Ocklenburg S, Schneider D, Burke M, Hengstler JG, Watzl C, Nitsche MA, Kumsta R, Wascher E, Genc E. Electrophysiological resting-state signatures link polygenic scores to general intelligence. Sci Rep. 2025 Nov 21;15(1):41170. doi: 10.1038/s41598-025-26778-4. PMID 41272243
- [Derived] Gajewski PD, Brode P, Claus M, Golka K, Hengstler JG, Reinders J, Watzl C, Wascher E, Getzmann S. Changes of cognitive functions and proinflammatory cytokines across the lifespan in latent Toxoplasma gondii infection. Brain Behav Immun Health. 2025 Sep 15;49:101105. doi: 10.1016/j.bbih.2025.101105. eCollection 2025 Nov. PMID 41018675
- [Derived] Gajewski PD, Brode P, Claus M, Golka K, Hengstler JG, Watzl C, Wascher E, Getzmann S. The association between hair cortisol and burnout is moderated by age, psychosocial, and immunological markers. Brain Behav Immun Health. 2024 Nov 23;43:100909. doi: 10.1016/j.bbih.2024.100909. eCollection 2025 Feb. PMID 39717874
- See also: This is the oficial site of the Dortmund Vital Study — https://vital-study.ifado.de/home